CLINICAL TRIAL: NCT04932109
Title: Development of a Subcutaneous Scar Scoring System Via Ultrasonography and Its Association With Hand Function in Traumatic Hand Injured Patients
Brief Title: Ultrasonographic Subcutaneous Scar Scoring System for Traumatic Hand Injured Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-ER-109-425
Record Dates: First submitted 2021-06-14; First posted 2021-06-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-01

CONDITIONS: Hand Injuries
Keywords: Traumatic hand injury; Ultrasonography; Subcutaneous scar
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Group
  Interventions: Other: No intervention
- Hand Injuries Group
  Interventions: Other: No intervention
- Healthcare professional: Clinical healthcare professionals who specialized in orthopedic, rehabilitation, hand anatomy, musculoskeletal ultrasound and so on
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention in this group

SUMMARY:
This study aims to develop an objective scar scoring system via ultrasonography and try to apply it to clinical using.

This study was divided into two parts. The first part of the study is an observational study design. The scar scoring system will be developed, and its test-retest reliability and criterion-related validity will be tested in this part.

The second part is also an observational study design. The clinical application of the system on traumatic injured patients is conducted in the second part. The results from this scar scoring system are correlated with hand function measurements. Moreover, every scar will be recorded three times within one month during routine rehabilitation to investigate the change.

ELIGIBILITY:
Inclusion Criteria:

* Above 20 years old
* Traumatic hand injury (distal from wrist joint above 8 weeks and within one year)
* Able to do active motion and resistive activities
* Understand and cooperate the experiment

Exclusion Criteria:

* Injured by burn
* Have impairment in peripheral nerve and affect the movement
* Combined with other central nerve deficits

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with traumatic hand injuries will be recruited from the Department of Rehabilitation in National Cheng Kung University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2024-11-26 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasonography platform - Healthy Group - Baseline | Baseline, 2 days after baseline
  An ultrasonography platform and different installed modes will be used to gather the images from dominant hand of healthy adults. These data will be collected two times in healthy group to test the test-retest reliability of the system.
Ultrasonography platform - Healthy Group - 2 days after baseline | Baseline, 2 days after baseline
  An ultrasonography platform and different installed modes will be used to gather the images from dominant hand of healthy adults. These data will be collected two times in healthy group to test the test-retest reliability of the system.
Ultrasonography platform - Hand Injuries Group - Baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  An ultrasonography platform and different installed modes will be used to gather the images from affected and unaffected hand of patients with hand injuries. These data will be collected three times in hand injuries group to know how will the tissue change between different time points.
Ultrasonography platform - Hand Injuries Group - 2 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  An ultrasonography platform and different installed modes will be used to gather the images from affected and unaffected hand of patients with hand injuries. These data will be collected three times in hand injuries group to know how will the tissue change between different time points.
Ultrasonography platform - Hand Injuries Group - 4 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  An ultrasonography platform and different installed modes will be used to gather the images from affected and unaffected hand of patients with hand injuries. These data will be collected three times in hand injuries group to know how will the tissue change between different time points.
Goniometer - Hand Injuries Group - Baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The goniometer will be used to measure the range of motion (ROM) in the affected and affected finger.
Goniometer - Hand Injuries Group - 2 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The goniometer will be used to measure the range of motion (ROM) in the affected and affected finger.
Goniometer - Hand Injuries Group - 4 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The goniometer will be used to measure the range of motion (ROM) in the affected and affected finger.
Force sensors - Hand Injuries Group - Baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  A force sensor will be used to collect the single digit force data in affected and unaffected finger.
Force sensors - Hand Injuries Group - 2 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  A force sensor will be used to collect the single digit force data in affected and unaffected finger.
Force sensors - Hand Injuries Group - 4 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  A force sensor will be used to collect the single digit force data in affected and unaffected finger.
Hand dynamometer - Hand Injuries Group - Baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  Hand dynamometer will be used to measure the grip strength and pinch strength.
Hand dynamometer - Hand Injuries Group - 2 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  Hand dynamometer will be used to measure the grip strength and pinch strength.
Hand dynamometer - Hand Injuries Group - 4 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  Hand dynamometer will be used to measure the grip strength and pinch strength.
Purdue pegboard test - Hand Injuries Group - Baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The Purdue pegboard test will be used to test the unimanual and bimanual manipulation versus hand dexterity.
Purdue pegboard test - Hand Injuries Group - 2 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The Purdue pegboard test will be used to test the unimanual and bimanual manipulation versus hand dexterity.
Purdue pegboard test - Hand Injuries Group - 4 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The Purdue pegboard test will be used to test the unimanual and bimanual manipulation versus hand dexterity.
Disabilities of the Arm, Shoulder and Hand - Hand Injuries Group - Baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The Disabilities of the Arm, Shoulder and Hand (DASH) is a questionnaire, which will be used to evaluate disorders and measure disability of the upper extremities and monitor change or function over time.
Disabilities of the Arm, Shoulder and Hand - Hand Injuries Group - 2 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The Disabilities of the Arm, Shoulder and Hand (DASH) is a questionnaire, which will be used to evaluate disorders and measure disability of the upper extremities and monitor change or function over time.
Disabilities of the Arm, Shoulder and Hand - Hand Injuries Group - 4 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The Disabilities of the Arm, Shoulder and Hand (DASH) is a questionnaire, which will be used to evaluate disorders and measure disability of the upper extremities and monitor change or function over time.
Ultrasonography platform - Healthcare professional - Baseline | Baseline, within 1 week after baseline
  An ultrasonography platform and different installed modes will be used to gather the images. The healthcare professionals will as the users to collect images from phantom or hand tissues. These data will be collected up to two times in healthcare professional group to test the test-retest reliability of the system and the effect of different experience levels.
Ultrasonography platform - Healthcare professional - within 1 week after baseline | Baseline, within 1 week after baseline
  An ultrasonography platform and different installed modes will be used to gather the images. The healthcare professionals will as the users to collect images from phantom or hand tissues. These data will be collected up to two times in healthcare professional group to test the test-retest reliability of the system and the effect of different experience levels.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan